CLINICAL TRIAL: NCT03638934
Title: Efficacy of Decision Aid for Advanced Care Planning(RCT) for General Population: Randomized Controlled Trial
Brief Title: Efficacy of Self-education Program for Advanced Care Planning(RCT) for General Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Institute of Health, Korea (Other Government); National Clinical Research Coordination Center, Seoul, Korea (Other Government); National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Principal Investigator, Young Ho Yun, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HC15C1391-4
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Advance care planning

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videos about ACP (Experimental): Subjects in experimental group get three videos about advanced care planning based on Smart Management Strategy for Health (SMASH). After they finish watching the materials, they fill out the questionnaire.
  Interventions: Other: Videos about ACP
- Brochure for Life-Sustaining Treatment (Active Comparator): Subjects in the group get 13-page brochure entitled, Understanding the Life-Sustaining Treatment Act. After they finish watching the materials, they fill out the questionnaire.
  Interventions: Other: Brochure about Life-Sustaining Treatment Act

INTERVENTIONS:
Other: Videos about ACP — Three videos about advanced care planning are provided for self-education.
  Arms: Videos about ACP
Other: Brochure about Life-Sustaining Treatment Act — Brochure about Life-Sustaining Treatment Act are provided for self-education.
  Arms: Brochure for Life-Sustaining Treatment

SUMMARY:
This study verifies efficacy of Self-education program for advanced care planning in general population. Half of participants will receive a 20 minutes video about advanced care planning while the other half will receive a 13-page brochure entitled, Understanding the Life-Sustaining Treatment Act.

DETAILED DESCRIPTION:
This study validates effectiveness of decision aid that the investigators developed due to the rates of completing Advanced care planning are considerably low, which is led by the lack of information available to general population; whether they elevate the preference of healthy general population toward Advanced Care planning, reduce the burden of decision making, and support general population to overcome their crisis, compare to educational resources that are currently available.

Previous studies inform that educational video about advanced care planning increases the knowledge of care for life prolongation and affects the preference towards care for life prolongation and palliative care. However, previous studies focused mainly on patient populations, and the general population might differ in its understanding of disease, health care services, and ACP. In this study, we constructed ACP video decision support materials for the general population and compared their effectiveness in an RCT.

Primary outcome of this study is attitude and behavior change toward advanced care planning. Participants of this study will fill out the baseline questionnaire about ACP preference, end-of-life care preference, knowledge of ACP, etc. After that, participants will be allocated equally into the intervention group and the control group. Participants assigned to the intervention arm viewed the 20-minute educational decision support video entitled Advance Care Planning, which had been used and tested in studies with advanced cancer patients. Participants randomized to the attention-control arm received and read a 13-page brochure entitled, Understanding the Life-Sustaining Treatment Act, which was developed by the Ministry of Health and Welfare. After reading and watching the educational materials, patients will get another questionnaire about knowledge of ACP, satisfaction on the materials, ACP Preference, etc.

ELIGIBILITY:
Inclusion Criteria:

* Subject 20 years old and more
* Subject who understands the purpose of the study and signs with informed consent form

Exclusion Criteria:

* Inability to speak, understand, or write Korean
* Inability to understand the contents of the provided materials due to poor eyesight and hearing

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Changes in Advance Care Preference | Baseline, within 1 week
  Comparison the result of Advance Care Preference questionnaire

SECONDARY OUTCOMES:
Changes in Hospital Anxiety and Depression Scale | Baseline, within 1 week
  Comparison the result of Hospital Anxiety and Depression Scale questionnaire
Changes in CPR knowledge | Baseline, within 1 week
  Comparison the result of Changes in CPR knowledge questionnaire
Changes in palliative care / advance care planning knowledge score | Baseline, within 1 week
  Comparison the result of Changes in palliative care / advance care planning knowledge score questionnaire
Changes in No CPR preference in terminal status | Baseline, within 1 week
  Comparison the result of No CPR preference in terminal status questionnaire
Changes in End-of-Life care | Baseline, within 1 week
  Comparison the result of End-of-Life care preference questionnaire
Satisfaction on educational materials | Baseline, within 1 week
  The result of Satisfaction on educational materials questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Young Ho Yun, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided